CLINICAL TRIAL: NCT03169088
Title: "Cook to Health 2" : Monitoring Wellbeing and Health in the Community
Brief Title: "Cook to Health Study 2 ": Monitoring Wellbeing and Health in the Community (Main Study)
Acronym: C2H2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC16.283
Record Dates: First submitted 2017-04-11; First posted 2017-05-30 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: eating Behavior; Volunteers
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching procedure (Experimental): Volunteers will received Updated National Dietary Guidelines about food and physical activity with a one-year follow-up, plus connected coaching.
  Interventions: Other: Coaching procedure

INTERVENTIONS:
Other: Coaching procedure — In this study, the volunteers will be followed during one year.
  The wellbeing will be followed with :
  * survey like FFQ, IPAQ, SF36, dietary habits.
  * actimetry measurement
  * one year follow-up of weight, waist measurement
  * nutritional biomarkers

SUMMARY:
Unhealthy lifestyles are major factors contributing to chronic conditions that impose a huge financial burden in EU healthcare systems. Unfortunately, the communication of Public Health failed to influence consumer to change their habits.

In this study, the aim is to evaluate the impact of a regular monitoring during 1 year on wellbeing and dietary habits in healthy volunteers.

This study follows the pilot study "cook to health" and is intended to confirm the results obtained by the tools used in C2H, in a larger population (25-50 years)

DETAILED DESCRIPTION:
Today, medicine mainly curative and reactive is primarily interested in sick people. Now, with our aging Western populations, we face a strong increase in chronic diseases incidence / prevalence that have a financial cost that becomes unbearable. Society's resources are being drained by the rising costs of disease management and of incremental improvements to our existing health care system. Immediate action is required to reverse these trends. The paradigm shift would be to move from a reactive to a proactive medicine that promote healthy life style to decrease incidence of chronic conditions through P4 Medecine that is Preventive, Participative, Predicitive and Personnalized.

However, unhealthy lifestyles are major factors contributing to chronic conditions that impose a huge financial burden in EU healthcare systems. Insufficient physical activity, poor diet and obesity are significant risk factors for cancers, cardiovascular, chest, metabolic disorders and leading causes of morbidity and premature mortality. Clinically studies indicate that different conditions can be prevented and sometimes reversed through adaptation of healthy habits. But the communication of Public Health failed to influence consumer to change their habits. Hence, it is recognized as a gold standard that better nutrition and better health will reduce the risk of chronic diseases such as obesity and cardiovascular diseases, which impact heavily on health spending. A report by the French National Assembly estimated the cost of obesity for the health insurance, if we add the daily allowances of sick care costs, between 2 and 6 € billion / year (until 4.6% of current health expenditure). As recently summarized by Caroline K. Kramer I 2015 moderate weight loss is related to favorable clinical outcomes. A weight loss of 7% (modification of lifestyle) reduced diabetes progression (-58%). The data collected addressed to health professionals will also enable better guide diagnostics and more efficient care strategies. Unfortunately free-living individuals are often poor at judging the healthiness of their own diet (choice of meal constituents, cooking methods, and portion sizes pattern of eating). Moreover, there is a lack of awareness of the contextual features influencing eating behavior and even where there is motivation to change, people have difficulty translating good intentions into healthy behaviors. Hence, their day-to-day constraints (lack of time, lack of knowledge, constraining family and cultural habits, personal tastes) make it difficult for them to comply and adopt the nationally recommended healthy lifestyles.

In this study, the volunteers will be followed during one year.

The wellbeing will be followed with :

* survey like FFQ, IPAQ, SF36, dietary habits.
* actimetry measurement
* one year follow-up of weight, waist measurement
* nutritional biomarkers

ELIGIBILITY:
Main Inclusion Criteria:

* 25 y ≤ Age ≤50 y
* Live in a family and be the main person who prepares meals
* Be able to use the personal health monitoring devices;
* Consenting adults based in Grenoble area France
* have a valid Internet connection with access from home;
* Be legally able to give consent.
* Person affiliated to social security

Main Exclusion Criteria:

* Be under chronic use of medications; (except contraception or chronic treatment for headache)
* Vital prognosis engaged within 12 months;
* Recent surgical intervention or hospitalization (< 6 months)
* Being unable to understand, follow objectives and methods due to cognition or language problems;
* Be likely to move away from the geographic inclusion zone (mainland France);
* Be unavailable (e.g. work commitment abroad) for the two months following inclusion;
* Pregnant women, feeding and parturient
* Playing sports at a high level (more than 7h/week our 1h/day)
* Subject under administrative or judicial control, person who are protected under the act.
* Daily alcohol consumption >20g for women and > 30g for men

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Alternate Healthy Eating Index-2010 (AHEI-2010) score | 1 year
  calculated by Food Frequency Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PISON, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hood L, Auffray C. Participatory medicine: a driving force for revolutionizing healthcare. Genome Med. 2013 Dec 23;5(12):110. doi: 10.1186/gm514. eCollection 2013. No abstract available. PMID 24360023
- [Background] Hood L, Flores M. A personal view on systems medicine and the emergence of proactive P4 medicine: predictive, preventive, personalized and participatory. N Biotechnol. 2012 Sep 15;29(6):613-24. doi: 10.1016/j.nbt.2012.03.004. Epub 2012 Mar 18. PMID 22450380
- [Background] Hood L, Price ND. Demystifying disease, democratizing health care. Sci Transl Med. 2014 Feb 26;6(225):225ed5. doi: 10.1126/scitranslmed.3008665. No abstract available. PMID 24574336
- [Background] Dzau VJ, Ginsburg GS, Van Nuys K, Agus D, Goldman D. Aligning incentives to fulfil the promise of personalised medicine. Lancet. 2015 May 23;385(9982):2118-9. doi: 10.1016/S0140-6736(15)60722-X. Epub 2015 May 6. No abstract available. PMID 25957453
- [Background] Kramer CK. Weight loss is a useful therapeutic objective. Can J Cardiol. 2015 Feb;31(2):211-5. doi: 10.1016/j.cjca.2014.08.003. Epub 2014 Aug 14. PMID 25661556
- [Background] Scalbert A, Brennan L, Manach C, Andres-Lacueva C, Dragsted LO, Draper J, Rappaport SM, van der Hooft JJ, Wishart DS. The food metabolome: a window over dietary exposure. Am J Clin Nutr. 2014 Jun;99(6):1286-308. doi: 10.3945/ajcn.113.076133. Epub 2014 Apr 23. PMID 24760973
- [Background] Chiuve SE, Fung TT, Rimm EB, Hu FB, McCullough ML, Wang M, Stampfer MJ, Willett WC. Alternative dietary indices both strongly predict risk of chronic disease. J Nutr. 2012 Jun;142(6):1009-18. doi: 10.3945/jn.111.157222. Epub 2012 Apr 18. PMID 22513989
- [Background] Gooding HC, Shay CM, Ning H, Gillman MW, Chiuve SE, Reis JP, Allen NB, Lloyd-Jones DM. Optimal Lifestyle Components in Young Adulthood Are Associated With Maintaining the Ideal Cardiovascular Health Profile Into Middle Age. J Am Heart Assoc. 2015 Oct 29;4(11):e002048. doi: 10.1161/JAHA.115.002048. PMID 26514160
- [Derived] Castellano-Escuder P, Gonzalez-Dominguez R, Vaillant MF, Casas-Agustench P, Hidalgo-Liberona N, Estanyol-Torres N, Wilson T, Beckmann M, Lloyd AJ, Oberli M, Moinard C, Pison C, Borel JC, Joyeux-Faure M, Sicard M, Artemova S, Terrisse H, Dancer P, Draper J, Sanchez-Pla A, Andres-Lacueva C. Assessing Adherence to Healthy Dietary Habits Through the Urinary Food Metabolome: Results From a European Two-Center Study. Front Nutr. 2022 Jun 9;9:880770. doi: 10.3389/fnut.2022.880770. eCollection 2022. PMID 35757242